CLINICAL TRIAL: NCT04538963
Title: Arrest of Proximal Caries Using Orthodontic Bands and Glass Ionomer Cement as a Preventative Intervention: A Split Mouth Study
Brief Title: Arrest of Proximal Caries Using Orthodontic Bands and Glass Ionomer Cement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Macaire Thiel, Principal Investigator, Pediatric Dentist, Medical College of Wisconsin
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 1554245
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Dental Caries Class II; Dental Caries in Children; Dental Caries on Smooth Surface Limited to Enamel

STUDY DESIGN:
Intervention Model Description: Split-mouth design- individual patient has a pair of carious lesions; one will receive the intervention, the other will be monitored per standard of care.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor (individual assessing radiographs for evidence of carious lesion progression or stabilization) will be masked. Due to the nature of the intervention (orthodontic band placement), the participant and care providers will not be able to be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Banded Tooth (Experimental): This tooth will have an orthodontic band and glass ionomer cement placed as an intervention for interproximal incipient caries.
  Interventions: Device: Orthodontic Band affixed with Glass Ionomer Cement
- Non-banded Tooth (No Intervention): This tooth will be monitored per standard of care; encourage good dental hygiene at home.

INTERVENTIONS:
Device: Orthodontic Band affixed with Glass Ionomer Cement — Glass ionomer cement utilized to affix a blank orthodontic band to the tooth; the mechanical retention of the band will also help retain cement in contact with the tooth- the hypothesis is that the fluoride release from the cement will aid in remineralization of tooth structure.
  Arms: Banded Tooth

SUMMARY:
The purpose of this study is to evaluate the efficacy of using orthodontic bands with glass ionomer cement to arrest or reverse interproximal lesions as a preventive treatment compared to monitoring and oral hygiene.

The investigators hypothesize that placing orthodontic bands with glass ionomer cement will arrest and possibly remineralize incipient carious lesions compared to teeth that are being monitored without intervention.

DETAILED DESCRIPTION:
This study is designed to determine the efficacy of orthodontic bands and glass ionomer cement in arresting and remineralizing incipient carious lesions as compared to monitoring for changes.

This is a single blinded, split mouth randomized control trial, with the patient being their own control. A split mouth study is considered the gold standard because both experimental and control groups are exposed to the same environmet and conditions within the mouth. This study design eliminates confounding variables that may occur that could significantly alter the interpretation of end results (e.g. oral hygiene effectiveness between two patients).

Participants will be screened at their routine periodic dental examination, where they will receive a dental exam, prophylaxis (cleaning), radiographs and fluoride varnish application in accordance with the guidelines from the American Academy of Pediatric Dentistry. Radiographs will be examined by an evaluator to determine if participants meet the inclusion criteria. Each participant requires at least one pair of permanent posterior teeth with interproximal caries lesions in enamel or in proximity of the dentinal enamel junction (E1, E2, early D1). An ideal pair consists of the same tooth type on the left and right side of the mouth (i.e. tooth #5 and #12, maxillary right permanent first premolar and maxillary left permanent first premolar). Another acceptable type of pair is same tooth type (i.e. tooth #5 and #21, maxillary right permanent first premolar and mandibular left permanent first premolar) or two adjacent teeth (i.e tooth #19 and 18 mandibular left first and second molar). Additionally, patients may also be screened when coming in for other dental treatment as well.

Each participant will have his or her qualifying lesions randomized equally into two groups, one that will receive the band, and one that will not. Envelopes will contain the treatment conditions: Left/Upper/Distal or Right/Lower/Mesial, to indicate that the lesion on either the left/upper/distal or right/lower/mesial side of the mouth will get banded. They will be randomly organized and then ordered in the box.

After randomization has occurred, each participant will have a blank orthodontic band (Denovo) fitted on the treatment lesion and cemented with glass ionomer cement (Fuji). Additionally, oral hygiene instructions will be reinforced. Participants will be instructed to return for their routine periodic dental exam in 6 months. Because the intervention is obvious, blinding the patient or the operator is not possible. At the 6 month visit, the band will be removed with a band remover prior to their dental exam and cleaning. Routine radiographs (according to the AAPD's radiographic guidelines) will be taken after the band has been removed. 20,21,22

A blinded second investigator will examine the pre and post treatment radiographs. Lesions will be classified initially by ADA CCS, and change will be noted as: progression, arrest, or regression. A de-identified data sheet containing the data will be sent to a statistician and a McNemar's Chi-square test will be used to test the differences in the lesion status of both groups

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Children or adolescents (Age 5<17.5yrs) who have erupted permanent teeth that make interproximal contact with other teeth, either primary or permanent teeth.
* Presence of at least one pair of interproximal carious lesions (E1, E2, early D1 according to the ADA CCS), evaluated by radiographic analysis, on permanent premolars or molars that do not require surgical intervention. If multiple pairs of lesions are present, they may be included in the study as well.

Exclusion criteria

* Patients who will be undergoing orthodontic treatment in the following 12 months.
* Patients with a poor behavior rating at their dental visit, defined with a (--) designation in behavior note
* Patients noted to have severe plaque levels and generalized severe gingivitis.
* Teeth with advanced caries into dentin that require surgical intervention restoration (Mid D1-D3). Dental needs that are required will be completed by the primary dental provider in the Dental Clinic

Ages: 5 Years to 209 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Radiographic Assessment of Interproximal Carious lesions | 6 months from previous recall visit
  Review of radiographs to assess if carious lesions have progressed or stabilized over time

CONTACTS AND LOCATIONS:
Overall Officials: Macaire C Thiel, DDS MS, Principal Investigator — Children's Hospital of Wisconsin, Pediatric Dental Residency Program Faculty
Locations (2):
- United States (2):
  - Children's Dental Center- Downtown, Milwaukee, Wisconsin
  - Children's Dental Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No